CLINICAL TRIAL: NCT03716778
Title: Enhanced Effectiveness of Combined Eccentric and Concentric Exercise Over Traditional Cardiac Exercise Rehabilitation Program in Patients With Chronic Heart Failure: a Randomized Controlled Study
Brief Title: Rehabilitation by Eccentric Exercise in Heart Failure Patients
Acronym: REX-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This premature end of the study is due to the lack of human resources and the fact that the forceps used to perform the biopsies for this study have not been marketed since January 2023.
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Clinique Médicale Cardio-Pneumologique de Durtol (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-411; 2017-A00969-44 (Other: 2017-A00969-44)
Record Dates: First submitted 2018-10-08; First posted 2018-10-23 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Chronic Heart Failure Patient; Rehabilitation Program
Keywords: Heart failure; eccentric; exercise; rehabilitation program; exercise testing; 6 min. walk test
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical exercise training modality in concentric mode (CON) (Other): Description: Control group, usual medical care according to the rehabilitation recommendations
  Interventions: Other: Eccentric rehabilitation sessions
- experimental, active group (ECC) (Experimental): Patients perform a mixed program combining eccentric pedalling session with the usual sessions
  Interventions: Other: Eccentric rehabilitation sessions

INTERVENTIONS:
Other: Eccentric rehabilitation sessions — ECC cycling will be conducted using a commercially available ECC motor-driven ergometer. Intensity and duration are progressively increased during the first five sessions in order to minimize the extent of exercise-induced muscle soreness.
  The subjects will perform five sessions of endurance training on cycle ergometer per week. Each session lasting 30 minutes will be achieved at an intensity corresponding to the pre-determined CON ventilatory threshold. In the ECC group, 3 sessions of ECC (Monday, Wednesday and Friday) and two session of concentric (Tuesday and Thursday) cycling will be carried out each week. In the control group CON all sessions will be achieved using the traditional pedaling mode.

SUMMARY:
As part of the regular rehabilitation program for chronic heart failure (CHF) patients, the addition of dynamic eccentric endurance (ECC) exercise sessions to the conventional concentric cycling program (CON) would enable greater gains in functional capacity that the CON alone. Furthermore, in the case of severe heart failure, results of conventional exercise rehabilitation remains limited on account of the poor physical fitness and deconditioning. Dynamic ECC has been shown to enhance muscle mass and improve muscle strength in subjects with functional limitations comparable to those in CHF, but to date reports on effects on muscle endurance and overall functional capacity remain scarce or non-existent.

Investigator hypothesize that a combination of these two types of training will allow both an improvement in strength and oxidative muscle capacities. These benefits must be objectified at the level of the walking distance covered in 6 min (6-WT).

DETAILED DESCRIPTION:
Investigator hypothesize that the combination of CON and ECC forms of endurance exercise will potentiate peripheral muscle and cardio-circulatory adaptations. All sessions, regardless of the modality, will be performed at the same percentage of the concentric peakVO2. Sessions performed in ECC mode will induce a mechanical overload. The ECC training of such intensity and duration seemingly having little or no effect on mitochondrial muscle adaptations, the maintenance of conventional training will allow stimulation of the aerobic endurance component. A synergistic effect is expected from the combination of the two modalities; the muscle strength gain induced by ECC allowing to sustained greater cycling workloads yet compatible with the cardio-circulatory capabilities of patients with CHF and more specifically their exercise cardiac output adjustment.

Investigator chose to assess the extent of benefits through functional capacity tests reflecting adaptation of both the aerobic (endurance capacity) and anaerobic (muscle strength) components of adaptive response, namely, 1) 6 min. walk test (6-WT), 2) time up and go test (TUGT), 3) quadriceps isometric muscular strength (IMS) and gait speed test.

The study is a prospective, open, controlled and randomized study in two parallel groups carried out in a single center. Patients will be included in the study if: i) they are referred to the cardiac rehabilitation center for the 5-week training program, ii) they meet the inclusion criteria and iii) they provide their signed consent.

Patients will be followed for 5 weeks, the duration of the cardiac rehabilitation program. They will benefit from the standard evaluation of any CHF patient referred for rehabilitation including an initial 12-lead ECG, a trans-thoracic cardiac ultrasound assessment and a cycling exercise stress test with gas exchange analysis and non-invasive measurement of cardiac output using a bio-impedance device. A standard biological blood analysis will be performed for NFS-platelets, blood electrolytes, CRP, NTproBNP, nutritional status with albumin and pre-albumin.

All subjects will perform 5 exercise sessions per week on a cycle ergometer. As per randomization outcome, the "intervention" group will perform three of the five weekly sessions in ECC mode (the other two in CON) while the control group will perform the five weekly sessions in CON mode.

The intensity of the cycling will be the same in both groups as determined from the initial cycling incremental test targeted to correspond to the VO2 associated with the ventilatory threshold.

ELIGIBILITY:
Inclusion Criteria:

* Patient with systolic chronic heart failure
* Patients aged 18 to 75 years
* Referred for participation in the 5-week rehabilitation program
* At a time distance from an acute coronary syndrome or myocarditis (less than 3 months old) and clinically stabilized.
* Beneficiary or affiliated with social security coverage

Exclusion Criteria:

* All the usual criteria considered contra-indicated for cardiac exercise rehabilitation according to the consensus recommendations ( REF)
* Non-stabilized acute coronary syndrome
* Decompensated heart insufficiency
* Stage IV NYHA
* Severe, uncontrolled disturbances in ventricular rhythm
* Presence of an intracardiac thrombus with high risk of embolism
* Presence of pericardial effusion of medium to high importance
* Recent history of thrombophlebitis with or without pulmonary embolism
* Obstacle to severe and / or symptomatic left ventricular ejection
* Any progressive inflammatory and / or infectious condition
* Severe and symptomatic pulmonary arterial hypertension
* Inability to perform physical activity
* Reversible heart disease
* Patients undergoing circulatory assistance
* Patients taking blood thinner medication (except Kardegic-type aggregates and direct oral anticoagulants)
* Patients with known allergy to Xylocaine
* Pregnant or lactating women
* Women of childbearing age without contraception
* Patient under tutorship, curatorship or deprived of liberty

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
6 min. walk test (6-WT) | at day 1
  6 min. walk test (6-WT)
6 min. walk test (6-WT) | at the end of the rehabilitation program (at the end of the 5 weeks)
  6 min. walk test (6-WT)

SECONDARY OUTCOMES:
Time up and go test (TUGT) | at day 1
  Test that evaluates seated transfers, standing, walking and changes of direction.
Time up and go test (TUGT) | at the end of the rehabilitation program (at the end of the 5 weeks)
  Test that evaluates seated transfers, standing, walking and changes of direction.
Quadriceps isometric muscular strength | at day 1
  The maximum muscle strength of the quadriceps (dominant limb) will be measured on a bench according to the instructions
Quadriceps isometric muscular strength | at the end of the rehabilitation program (at the end of the 5 weeks)
  The maximum muscle strength of the quadriceps (dominant limb) will be measured on a bench according to the instructions
Gait speed test | at day 1
  Test that evaluate walking speed over 4 meters
Gait speed test | at the end of the rehabilitation program (at the end of the 5 weeks)
  Test that evaluate walking speed over 4 meters
Results of the incremental tests | at day 1
  Peak VO2
Results of the incremental tests | at the end of the rehabilitation program (at the end of the 5 weeks)
  Peak VO2
Body composition measurements | at day 1
  fat body mass
Body composition measurements | at day 1
  lean body mass
Body composition measurements | at the end of the rehabilitation program (at the end of the 5 weeks)
  fat body mass
Body composition measurements | at the end of the rehabilitation program (at the end of the 5 weeks)
  lean body mass
Muscle Biopsie | at day 1
  mitochondrial and histo-biochemical functionality from muscle biopsies
Muscle Biopsie | at the end of the rehabilitation program (at the end of the 5 weeks)
  mitochondrial and histo-biochemical functionality from muscle biopsies
Metabolomic analysis | at day 1
  identification of specific blood and muscle biomarkers in response to retraining
Metabolomic analysis | at the end of the rehabilitation program (at the end of the 5 weeks)
  identification of specific blood and muscle biomarkers in response to retraining

CONTACTS AND LOCATIONS:
Overall Officials: Ruddy RICHARD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Plaquevent-Hostache G, Touron J, Costes F, Perrault H, Clerfond G, Cuenin C, Moisa A, Pereira B, Boiteux MC, Eschalier R, Richard R. Effectiveness of combined eccentric and concentric exercise over traditional cardiac exercise rehabilitation programme in patients with chronic heart failure: protocol for a randomised controlled study. BMJ Open. 2019 Sep 26;9(9):e028749. doi: 10.1136/bmjopen-2018-028749. PMID 31558450